CLINICAL TRIAL: NCT04889690
Title: A Multiple Ascending Dose Study To Assess Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of ACH-0144471 In Healthy Volunteers
Brief Title: Study of Multiple Doses of Danicopan in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ACH471-002
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Healthy
Keywords: Danicopan; ALXN2040; ACH-0144471; Factor D Inhibitor; Pharmacokinetics; Pharmacodynamics; Ascending Dose
MeSH Terms: interventions — danicopan; rhoA GTP-Binding Protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1: 200 mg (Experimental): All participants under fasted conditions received 200 mg of danicopan or placebo twice daily (BID) over a 14-day period.
  Interventions: Drug: Danicopan; Drug: Placebo
- Cohort 2: 500 mg (Experimental): All participants under fasted conditions received 500 mg of danicopan or placebo BID over a 14-day period.
  Interventions: Drug: Danicopan; Drug: Placebo
- Cohort 3: 800 mg (Experimental): All participants under fasted conditions received 800 mg of danicopan or placebo BID over a 14-day period.
  Interventions: Drug: Danicopan; Drug: Placebo
- Cohort 4: 75 mg (Experimental): All participants under fasted conditions received 75 mg of danicopan or placebo thrice daily (TID) over a 7-day period.
  Interventions: Drug: Danicopan; Drug: Placebo

INTERVENTIONS:
Drug: Danicopan
  Other Names: ACH-0144471 (formerly); ALXN2040; ACH-4471; ACH4471; 4471
Drug: Placebo

SUMMARY:
This was a multiple ascending dose, randomized, double-blind study assessing the safety, tolerability, pharmacokinetics, and pharmacodynamics of danicopan in healthy participants. Four different doses (75 milligrams [mg], 200 mg, 500 mg, 800 mg) and dose-matched placebo were administered under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy was defined as having no clinically relevant abnormalities identified by a detailed medical history, physical exam, blood pressure and heart rate measurements, 12-lead electrocardiogram, and clinical laboratory tests.
* Body mass index of 18 to 30 kilograms (kg)/meter squared with a minimum body weight of 50 kg.

Exclusion Criteria:

* History or clinically relevant evidence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
* Any condition possibly affecting drug absorption (including gastrectomy and cholecystectomy).
* Body temperature greater than or equal to 38°Celcius on Day -1 or Day 1, Hour 0; history of febrile illness or other evidence of infection within 14 days prior to first study drug administration.
* Current tobacco/nicotine user; consumption of any alcohol within 72 hours before first study drug administration or have a history of regular alcohol consumption exceeding 21 drinks/week within 6 months of screening; positive urine drug screen at screening or Day -1.
* Clinically significant laboratory abnormalities at either Screening or Day -1.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-05-21 (Actual); Primary Completion 2017-01-11 (Actual); Study Completion 2017-01-11 (Actual)

PRIMARY OUTCOMES:
Incidence Of Serious Adverse Events, Grade 3 Or 4 Adverse Events (AEs), AEs Leading To Discontinuation, And Clinically Significant Laboratory Abnormalities And Electrocardiogram Abnormalities | Day 1 through Day 42

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) Of Danicopan | Up to 16 hours postdose
Time To Maximum Observed Plasma Concentration (Tmax) Of Danicopan | Up to 16 hours postdose
Area Under The Plasma Concentration Versus Time Curve Over The Dosing Interval (AUCtau) Of Danicopan | Up to 16 hours postdose
Activity Of Danicopan As Measured By Alternative Pathway (AP) Wieslab Assay | Up to 16 hours postdose
Relationship Between AP Inhibition And Danicopan Plasma Concentrations | Up to 16 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No